CLINICAL TRIAL: NCT01594996
Title: A Multinational, Multicenter, Retrospective, Observational Drug Utilisation Study of Seroquel Extended Release (XR) Prescribed by Psychiatrists as Treatment for Major Depressive Disorder (MDD) in Selected Countries in the European Union (EU)
Brief Title: European Drug Utilization Study
Acronym: EUDUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1443C00057
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Seroquel XR; Quetiapine XR; Drug utilization; Major depressive disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Seroquel XR group

SUMMARY:
The purpose of this retrospective observational study is to evaluate the characteristics of patients receiving Seroquel XR as treatment for their Major Depressive Disorder. The study will also investigate how the medication is used for these patients and if there are any differences in drug utilisation between the included countries. The study is observing patients initiating Seroquel XR during a 9 month period corresponding to 3 to 12 months following the launch of the product in each country for the MDD indication. A drug utilisation questionnaire will be used to collect study data from patients' medical records.

DETAILED DESCRIPTION:
A Multinational, Multicenter, Retrospective, Observational Drug Utilisation Study of Seroquel Extended Release (XR) Prescribed by Psychiatrists as Treatment for Major Depressive Disorder (MDD) in Selected Countries in the European Union (EU)

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent before initiation of any collection of questionnaire data.
* Documented clinical diagnosis of Major Depressive Disorder, Single Episode, or Recurrent.
* Initiation of Seroquel XR for treatment of MDD during the period defining the inception cohort, i.e. from 3 months after launch until the index date (12 months after launch).

Exclusion Criteria:

* If participating in any clinical trial during the time from 3 months after launch until the index date, the patient cannot take part in this study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500-2000 patients that are broadly representative of the overall Major Depressive Disorder population in Europe. Patients are distributed at medical healthcare centres, private practice, as well as university and community hospitals in five European countries.
Sampling Method: Non-Probability Sample
Enrollment: 814 (Actual)
Dates: Start 2012-04-24 (Actual); Primary Completion 2014-03-27 (Actual); Study Completion 2014-03-27 (Actual)

PRIMARY OUTCOMES:
Patient age (mean and range) | Baseline
Patient gender (%) | Baseline
Diagnosis for which Seroquel XR was prescribed (% of Major Depressive Disorder- MDD) | Baseline
Patients hospitalized for any psychiatric condition (n, %) | follow-up up to nine months
Daily dose of Seroquel XR (mode and range) | follow-up up to nine months

SECONDARY OUTCOMES:
Patient referral pathway (%) | Baseline
Participating psychiatrist practice setting (%) | Baseline
Percent of patients experiencing psychotic symptoms at initiation of Seroquel XR (n, %) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hans A Eriksson, MD, Study Director — AstraZeneca R&D
Locations (1):
- Research Site, Dortmund, Germany

REFERENCES:
- See also: D1443C00057_Clinical_Study_Report_Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1761&filename=D1443C00057_Clinical_Study_Report_Synopsis.pdf
- See also: REDACTED_D1443C00057_Revised_NIS_Protocol_21-Jan-2016 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1761&filename=REDACTED_D1443C00057_Revised_NIS_Protocol_21-Jan-2016.pdf